CLINICAL TRIAL: NCT06883006
Title: RESET: Regulation of Emotion, Sleep Extension, and mTBI
Brief Title: Regulation of Emotion, Sleep Extension, and mTBI
Acronym: RESET
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merrimack College (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Laura Kurdziel, Associate Professor, Merrimack College
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB-FY18-19-196; 1R15MH136612-01A1 (NIH)
Record Dates: First submitted 2025-03-12; First posted 2025-03-19 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Brain Concussion; Brain Injuries, Traumatic; Sleep; Emotion Regulation
MeSH Terms: conditions — Brain Concussion; Brain Injuries, Traumatic; Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Extension (Experimental): A 1.5-hour nap opportunity compared to a neutral 1.5 hour waking activity (e.g., puzzle completion) prior to task. In this arm, participants will nap prior to the emotion regulation task. These two conditions will be counter-balanced within gender and participants will complete them 1 week apart. If they are in the nap condition, they will nap for 1.5 hours with PSG in a dark, soundproofed room with optional fan, white noise, or music.
  Interventions: Behavioral: Sleep Extension
- Wake Condition (No Intervention): A 1.5-hour nap opportunity compared to a neutral 1.5 hour waking activity (e.g., puzzle completion) prior to task. In this arm, participants will not nap prior to the emotion regulation task. These two conditions will be counter-balanced within gender and participants will complete them 1 week apart. If they are in the no nap condition, they will work on puzzles for 1.5 hours in the same room but with the lights on.

INTERVENTIONS:
Behavioral: Sleep Extension — A 1.5-hour nap opportunity compared to a neutral 1.5 hour waking activity (e.g., puzzle completion) prior to task. Participants will either nap or not prior to the emotion regulation task. These two conditions will be counter-balanced within gender and participants will complete them 1 week apart. If they are in the nap condition, they will nap for 1.5 hours with PSG in a dark, soundproofed room with optional fan, white noise, or music. If they are in the no nap condition, they will work on puzzles for 1.5 hours in the same room but with the lights on.
  Arms: Sleep Extension

SUMMARY:
Concussions are incredibly common, and often result in severe and long lasting symptoms, including, but not limited to, sleep deprivation and emotion dysregulation. This study aims to demonstrate the therapeutic benefits of sleep extension (napping) on emotion regulation in individuals after they sustain a concussion. Thus, sleep extension may be a cost-effective, low risk, supplemental treatment for those with emotion dysregulation following a concussion. The main questions it aims to answer are:

1. Is a nap an effective way to improve emotion regulation in individuals with a concussion?
2. Does a nap reduce the required executive resources necessary to regulate emotions in individuals with a concussion?

DETAILED DESCRIPTION:
The specific objective of this proposal is to determine whether sleep extension, in the form of a mid-day nap, improves emotion regulation in those with a mTBI, and to assess whether napping affects top-down neural control of emotion regulation. In order to test this, individuals with a recent (within ~1 month) mTBI (n=60) will complete an emotion regulation task after a nap (1.5 hour nap opportunity) and after a quiet wakefulness session (1.5 hour quiet waking bout). The nap will be recorded using polysomnography (PSG) to assess sleep stages and spectral analysis of sleep physiology. Emotion regulation will be assessed using a cognitive reappraisal task in which participants are asked to reduce their emotional arousal to negative images (e.g., picturing a different/happy outcome). During this task, pupillometry, eye movement behaviors (i.e., fixations and dwell times), event-related potentials (ERPs), and valence/arousal ratings will be measured. Participants will complete the task twice, one week apart, with order of the nap/no nap condition counterbalanced within gender. Thus, the investigators will have behavioral, neurophysiological, and self-report measures of emotion regulation. Sleep patterns and sleep quality data will be collected using sleep profiler headbands (to assess nocturnal sleep physiology prior to and following testing sessions), a wrist-worn actigraph and a sleep diary (to assess typical sleep patterns), polysomnography (to assess nap sleep physiology), and questionnaires. Participants will receive an actiwatch and a sleep profiler headband to wear beginning the day prior to their first laboratory session. The participant will wear the actiwatch through the day following the second session (9 days total), and will wear the sleep profiler headband on the night prior to and following each laboratory session (4 days total). Participants will also complete self-report questionnaires to report demographic information, overall sleep behaviors, current sleepiness, current positive and negative affect, and mTBI symptoms and history.

The investigators will examine the following specific aims: Aim 1: To determine the efficacy of a nap to improve emotion regulation in individuals with mTBI (n=60). Aim 2: To examine whether a nap reduces the required executive resources necessary to regulate emotions in individuals with mTBI (n=60). Exploratory Aim 1: To examine whether mid-day nap physiology correlates with emotion regulation. Exploratory Aim 2: To examine whether a mid-day nap impacts nocturnal sleep physiology.

This proposal impacts the field by seeking to shift the current clinical practice for mTBI, suggesting that naps may be a fruitful intervention for emotional symptoms and reduced sleep following mTBI. It will also be the first to examine the neurological impacts of a nap in individuals following mTBI and how it could alter emotion regulation. The findings of this R15 will be used to power a larger R01 clinical trial to examine the benefits of a multi-day nap protocol on emotion regulation in individuals with mTBI. The incorporation of naps into the therapeutic care for those with mTBI may have significant benefits to their emotional control and mental well-being. This would be a practical, cost-effective, and low risk supplemental treatment that could be used by any and all populations.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 35 years old.
2. Have normal or corrected to normal vision
3. Sustained a FIRST or SECOND concussion within the last 2-3 weeks
4. No sleep disorders
5. Is not a shift worker

Exclusion Criteria:

1. Under 18 or over 35 years old.
2. Not have corrected normal vision with glasses or contacts
3. Has an astigmatism in both eyes
4. Had a concussion over 3 weeks ago
5. Has sleep disorder
6. Is a shift worker

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation (Self-report) | Weeks 0 and 1
  After viewing each image, participants will rate the valence and arousal of the image by using the Self Assessment Manikin79 (SAM). Participants will also be asked how successful they were at following the instruction to maintain or reappraise their negative affect on a 1 to 4 scale.
Emotion Regulation (Behavioral measures) | Weeks 0 and 1
  The main eye tracking behaviors will focus on the area of interest (i.e., the most emotional portion of the image). For interest areas, the investigators will examine how often participants look directly within each area of interest ("fixations") and how long they look within each area of interest ("dwell time"). The investigators will also examine the proportion of interest area fixations and dwell time relative to the trial totals.
Executive Control over Emotions (Pupillometry) | Weeks 0 and 1
  Participants' pupil dilation, which indicates cognitive control beyond sympathetic activation, will be measured. Average pupil size (area; in mm) will be compared between various conditions to determine differences in top-down control of emotion regulation.
Executive Control over Emotions (Neurophysiology; ERP) | Weeks 0 and 1
  The cap, described below, will continue to be worn during the subsequent emotion regulation task to record event related potentials (ERP). The Late Positive Potential (LPP) is an ERP most observable in the midline, and occurs approximately 300 ms after the onset of a stimulus. LPP is associated with top-down control of emotion regulation.

SECONDARY OUTCOMES:
Sleep Duration and Sleep Patterns (Actigraphy) | Weeks 0-2
  Participants will wear an actigraph for 9 days (1 day prior to their first lab session until 1 day after their second lab session). The Actiwatch Spectrum (Philips Respironics, Inc., Bend, OR) that will be used in this study is a water-resistant, wrist-worn device with off-wrist detection and triaxial accelerometer to measure motion. Participants will wear the Actiwatch for the duration of the study. Actigraph data will be assessed for average total sleep time (TST), sleep onset variability, sleep offset variability, average sleep efficiency, detection of and variability of mid-day naps, as well as changes in nocturnal sleep duration and efficiency following a nap. Actigraphy will be used to control for variability in typical sleep behaviors, sleep quality, and sleep quantity across individuals.
Self-report Control measures | Weeks 0 and 1
  Participants will complete the PSQI, and the RPQ to assess sleep quantity/quality, and mTBI symptoms, respectively. They will also complete the PANAS and SSS to be used as covariates.
Self-report Control measures | Week 0
  Participants will report demographic information such as whether they have any neurological or sleep disorders and whether they are on any medications that could influence sleep and emotion regulation. These will be used as covariates.

OTHER OUTCOMES:
Sleep physiology (Polysomnography) | Weeks 0 and 1
  A 32-electrode cap (Easycap, Brain Products, GmbH, Germany) montage for polysomnographic recordings will be applied. This montage is sufficient for both EEG/ERP recordings, as well as for sleep scoring analysis according to the American Academy of Sleep Science. All nap PSG recordings will be analyzed using BrainVision Analyzer (Brain Products, GmbH, Germany). The cap montage will be worn during both the nap and no-nap bout.
Sleep physiology (Polysomnography) | Weeks 0-2
  The Advanced Brain Monitoring Sleep Profiler™ EEG Sleep Monitor headband will be used to record sleep physiology of the night prior to and the night after each laboratory session (4 nights total). The Sleep Profiler headbands use three frontopolar channels which provide EEG, EOG, and EMG signals to determine sleep staging (Sleep Profilers have been validated compared to PSG). The headbands will be applied by the participant and worn during nocturnal sleep in their typical home sleeping space.

CONTACTS AND LOCATIONS:
Locations (1):
- Merrimack College, North Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Public use and restricted access study data and associated documentation will be made available to the research community free of charge through the Discovery Informatics Platform for Research provided by Research Information Science & Computing (RISC) at the Brigham and Women's Hospital data repository hosted at National Sleep Research Resource (NSRR). De-identified individual-level data will be uploaded every six months, as required by NIMH, to NSRR, including after the first six months if applicable. However, primary aims data (e.g., behavioral data) will be hidden from public view until publication or one year after the end of the award period, whichever comes first.
Time Frame: De-identified individual-level data will be uploaded every six months, as required by NIMH, to NSRR, including after the first six months if applicable. However, primary aims data (e.g., behavioral data) will be hidden from public view until publication or one year after the end of the award period, whichever comes first.
Access Criteria: All de-identified study data that are not designated as restricted use will be made available as public use data to the research community via NSRR. Users of the public use data must register with NSRR and agree to the Terms of Use, which state, "Access to the resources is controlled by per-dataset-access control, and access is only granted to individuals who have completed the web-based Data Access and Use Agreement (DAUA). Each DAUA submission is reviewed by the NSRR Review Committee, and reviewers ascertain that use of data appears appropriate with the intention of data collected and that there is a commitment to keep the data stored securely by the end-user. NSRR DAUAs expire 3 years from the date access is granted and can be renewed by either submitting a new request for data access or by requesting an extension of the agreement in writing to the NSRR Review Committee" (NSRR website). Data users also agree not to share or redistribute any data downloads.
URL: https://sleepdata.org/